CLINICAL TRIAL: NCT00567762
Title: A Randomized, Placebo-controlled, Double-masked Study of 0.1% Tacrolimus(FK506) Ophthalmic Suspension in Vernal Keratoconjunctivitis
Brief Title: Phase III Study of 0.1% Tacrolimus(FK506) Ophthalmic Suspension in Patients With Vernal Keratoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FJ-506D-AC09
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Keratoconjunctivitis; Conjunctivitis
Keywords: Keratoconjunctivitis; vernal keratoconjunctivitis; FK506; Tacrolimus
MeSH Terms: conditions — Keratoconjunctivitis; Conjunctivitis; Conjunctivitis, Allergic | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): FK506 ophthalmic suspension
  Interventions: Drug: FK506
- 2 (Placebo Comparator): Base of eye drops
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: FK506 — Opthalmic suspension
  Other Names: tacrolimius
  Arms: 1
Drug: placebo — placebo eye drops
  Arms: 2

SUMMARY:
To investigate the efficacy and safety of FK506 ophthalmic suspension on eye symptoms in patients with vernal keratoconjunctivitis

DETAILED DESCRIPTION:
0.1% FK506 ophthalmic suspension were administered twice-a-day to patients with vernal keratoconjunctivitis in whom treatment with topical anti-allergic agents had been ineffective. The primary efficacy endpoint was the mean change from the baseline (before the treatment)in total score for objective clinical signs at the final observation. The safety of FK506 ophthalmic suspension was also investigated.

ELIGIBILITY:
Inclusion Criteria:

* Vernal keratoconjunctivitis patients diagnosed by "Guideline of diagnosis and treatment of allergic conjunctival disease"
* Patients with type I reactions defined by skin testing, antibody measurement, etc.
* Age over 6 years old

Exclusion Criteria:

* Subjects receiving systemic administration or subconjunctival injection of corticosteroid or immunosuppressants(ophthalmic and systemic medications) within 2-weeks of initiation of the study
* Subjects needed to wear contact lenses during treatment period on a testing eye
* Subjects complicating an eye infection

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-02; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Mean change from the baseline (before the treatment) in total score for objective clinical signs at the final observation | 4 weeks

SECONDARY OUTCOMES:
Mean change from the baseline in score for objective clinical signs and the score for each objective clinical sign | Week 1, 2 and 4
Subjective symptom score (Visual Analog Scale) | 4 weeks
The improvement rate of subjective symptoms | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Ehime
  - Hokkaido
  - Kagoshima
  - Kochi
  - Miyazaki
  - Osaka
  - Tochigi
  - Tokyo